CLINICAL TRIAL: NCT06688318
Title: Effectivity of Allogenic Umbilical Cord Mesenchymal Stem Cells Conditioned Media for Osteoarthritis of the Knee Joint: A Clinical Study of Functional Score and Magnetic Resonance Imaging Evaluation Using CartiGram
Brief Title: Effectivity of Allogenic Umbilical Cord Mesenchymal Stem Cells Conditioned Media for Osteoarthritis of the Knee Joint
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kementerian Riset dan Teknologi / Badan Riset dan Inovasi Nasional, Indonesia (Other Government)
Responsible Party: Principal Investigator, Bintang Soetjahjo, SpOT (K), MD. PhD, Kementerian Riset dan Teknologi / Badan Riset dan Inovasi Nasional, Indonesia, Kementerian Riset dan Teknologi / Badan Riset dan Inovasi Nasional, Indonesia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 932/VII/HREC/2024
Record Dates: First submitted 2024-11-11; First posted 2024-11-14 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Osteoarthritis Knee
Keywords: osteoarthritis knee; Mesenchymal Stem Cell; conditioned media
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OA Knee (Experimental): Knee Intraarticular Conditioned Media Injection
  Interventions: Biological: Intra-articular secretome injection therapy

INTERVENTIONS:
Biological: Intra-articular secretome injection therapy — Intra-articular secretome injection therapy from hypoxic umbilical cord mesenchymal stem cell conditioned media

SUMMARY:
Osteoarthritis (OA) is a joint disorder that often occurs and causes disability. This disorder is characterized by an inflammatory reaction in the synovial joints accompanied by a gradual degeneration process in the articular cartilage and sub-chondral bone. Current research has discovered that stem cells produce conditioned media (secretome, extra vesicles, and exosomes) that have tissue regeneration, immunomodulation, anti-inflammatory, and anti-apoptotic capabilities. Research on conditioned media for umbilical cord mesenchymal stem cells is still at the in vivo stage in experimental animals. For this reason, this study aims to conduct clinical experimental research (translational study) in patients with knee joint OA who were given umbilical cord mesenchymal stem cell conditioned media via intra-articular injection.

DETAILED DESCRIPTION:
The research was conducted as a clinical trial and translational study, involving a single group treated with intra-articular secretome injection therapy derived from hypoxic umbilical cord mesenchymal stem cell conditioned media.

This study explores the clinical application of conditioned media from umbilical cord mesenchymal stem cells for treating knee OA. Our preliminary clinical trial involves administering this conditioned media via intra-articular injections to patients, followed by assessments using functional scores and MRI with T2 mapping sequence. This approach aims to harness the therapeutic potential of MSC derivatives in a clinical setting, offering a novel and potentially less invasive alternative to conventional OA treatments. The aim of this study is to evaluate the effectiveness of intra-articular injections of conditioned media from umbilical cord mesenchymal stem cells in improving knee joint function and structural integrity in patients with osteoarthritis, as assessed by MRI and functional scoring.

ELIGIBILITY:
Inclusion Criteria:

* age over 45 years
* primary knee joint OA Kellgrance-Lawrence grade 2 or 3,
* never had surgery or intra-articular injection before,

Exclusion Criteria:

* currently experiencing local infections and/or systemic infections,
* have a history of autoimmune disorders or immunodeficiency,
* have had surgery or injections on the knee joint,

Min Age: 45 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2024-04-03 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Functional Score 1. Knee Injury and Osteoarthritis Outcome Score (KOOS), | 2,4,6 Months
  The Knee Injury and Osteoarthritis Outcome Score (KOOS) is a questionnaire designed to assess short and long-term patient-relevant outcomes following knee injury. The KOOS is self-administered and assesses five outcomes: pain, symptoms, activities of daily living, sport and recreation function, and knee-related quality of life.
  Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems as common in orthopaedic scales and generic measures. Scores between 0 and 100 represent the percentage of total possible score achieved.
Functional Score 2. Knee Society Score (KSS) | 2,4,6 Months
  The original KSS has a "Knee Score" section (7 items) and a "Functional Score" section (3 items). Both sections are scored from 0 to 100 with lower scores being indicative of worse knee conditions and higher scores being indicative of better knee conditions.
Functional Score 3. Western Ontario and McMaster Universities Arthritis Index (WOMAC) Score | 2,4,6 Months
  Higher scores indicate worse pain, stiffness, and functional limitations. The WOMAC measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68).

SECONDARY OUTCOMES:
Radiographic Evaluation | 2,4,6 Months
  Magnetic Resonance Imaging Evaluation using CartiGram

CONTACTS AND LOCATIONS:
Overall Officials: Bintang S Bintang Soetjahjo, MD, PhD, Principal Investigator — Dr. Moewardi Hospital
Locations (1):
- Moewardi General Hospital, Surakarta, Central, Indonesia

IPD SHARING:
Plan to Share IPD: No